CLINICAL TRIAL: NCT04644341
Title: Post Discharge Tele-monitoring of COVID-19 Survivors for Long-Term Impacts and Point-of-Care
Brief Title: Tele-monitoring of COVID-19 Survivors for Long-Term Impacts
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Function Four Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: B2020:114 (HS24395)
Record Dates: First submitted 2020-11-14; First posted 2020-11-25 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Blood Circulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID survivors: Individuals who were infected by CPVID-19 and recovered.
  Interventions: Combination Product: cardiovascular and respiratory systems monitoring

INTERVENTIONS:
Combination Product: cardiovascular and respiratory systems monitoring — only one group of individuals to observe the impact of COVID-19 on their cardiovascular and respiratory systems in long term.

SUMMARY:
To confront the COVID-19 pandemic hospitals need to maximize bed availability and minimize the duration of patients' stay as much as possible. Given the constraints, physicians are neither able to investigate the long-term effects of COVID-19 nor able to optimize extended treatments beyond the hospital. Physicians also do not have time to keep patients mobile and lucid during their hospital stays, resulting in longer recovery periods and further complications for patients. The investigators propose the development of a tele-monitoring solution for the long-term monitoring of COVID-19 survivors. Such a solution will help save significant healthcare costs by reducing the number of plausible future hospitalizations due to patient complications, providing valuable insights to various stakeholders from doctors to policymakers on the long-term effects of COVID-19, and improving patient care and treatment.

Using our team's existing bio-instrumentation technologies and years of experience, the investigators propose to develop a custom-designed miniaturized monitoring system capable of recording pulse oximetry (blood's oxygen level), blood pressure, heart rate and breathing and swallowing sounds. This solution will be non-invasive, easy to implement and will not require an assistant physically present. The system will be augmented by regular videoconferencing sessions with a medical practitioner. The frequency of the connection can be modified depending on the patient's condition and medical history in consultation with our team's physician.

By running the proposed project on a large scale, the expected outcomes will be: 1) collection of reliable and objective information on the long-term impacts of COVID-19, 2) developing an all-in-one technology for future applications, 3) collection of objective and actionable information that can be used to optimize care and treatment plans for patients, 4) better care and treatment for all strata of society regardless of the remoteness of the residence, and 5) improved mental health and recovery of patients.

DETAILED DESCRIPTION:
To confront the COVID-19 pandemic hospitals need to maximize bed availability and minimize the duration of patients' stay as much as possible. Given the constraints, physicians are neither able to investigate the long-term effects of COVID-19 nor able to optimize extended treatments beyond the hospital. Physicians also do not have time to keep patients mobile and lucid during their hospital stays, resulting in longer recovery periods and further complications for patients. The investigators propose the development of a tele-monitoring solution for the long-term monitoring of COVID-19 survivors. Such a solution will help save significant healthcare costs by reducing the number of plausible future hospitalizations due to patient complications, providing valuable insights to various stakeholders from doctors to policymakers on the long-term effects of COVID-19, and improving patient care and treatment.

Using our team's existing bio-instrumentation technologies and years of experience, the investigators will develop a custom-designed miniaturized monitoring system capable of recording pulse oximetry (blood's oxygen level), blood pressure, heart rate and breathing and swallowing sounds. This solution will be non-invasive, easy to implement and will not require an assistant physically present. The system will be augmented by regular videoconferencing sessions with a medical practitioner. The frequency of the connection can be modified depending on the patient's condition and medical history in consultation with our team's physician.

By running the proposed project on a large scale, the expected outcomes will be: 1) collection of reliable and objective information on the long-term impacts of COVID-19, 2) developing an all-in-one technology for future applications, 3) collection of objective and actionable information that can be used to optimize care and treatment plans for patients, 4) better care and treatment for all strata of society regardless of the remoteness of the residence, and 5) improved mental health and recovery of patients.

The goal of this project is to provide COVID-19 survivors a point-of-care facility by using an interactive virtual program to measure 4 main vital biological signals (blood pressure, heart rate, pulse oximetry, and respiratory sounds (that include both tracheal and lung breathing and swallowing sounds) and assess cognitive status of individuals remotely at their own home. The specific objectives are:

1. Assemble the existing and medically approved blood pressure and pulse oximetry miniaturized non-invasive devices along with a digital stethoscope, all to be connected to a smart phone operated by a custom-designed app to collect and store data on secure servers of the PI. One secure server is dedicated to the contact information of the patients and their unique codes, and another physically separate server is dedicated to patients' data after anonymizing.
2. Schedule videoconferencing sessions for a Research Assistant (RA) to interact with the patient regularly to help with recording the signals remotely and assess the cognitive and mood of the patients at their home.
3. Evaluate the above program on 20 COVID-19 patients for a period of 4 months.
4. Analyse the collected data during the 4 months observation period, and identify any consistent pattern of the long-term effect of COVID-19.
5. Disseminate the results in both scientific and public events, and plan future studies.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years,
* MoCA > 15
* Clinically diagnosed with COVID-19 and have had symptoms for a minimum of 5 days
* Must speak and understand English
* Must have wifi Internet and an smart phone

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals infected with COVID-19 with symptoms
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Change from baseline Systolic Blood Pressure at 4 months
  The change of systolic blood pressure from baseline
Breathing sounds average power | Change from normal range at baseline and at 4 months
  Average power of the breathing sounds within 100 to 500 Hz
Risk of aspiration | Change from normal range at baseline and at 4 months
  risk of aspiration calculated from swallowing and breathing sounds pattern
SaO2 level | Change from normal range at baseline and at 4 months
  SaO2 level measured by pulse Oximetry

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Change from normal range at baseline and at 4 months
  Cognitive assessment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Once we collect data and they are useful, we plan to share the anonymized data on our website after receiving Ethics Board's approval.